CLINICAL TRIAL: NCT02637791
Title: A Low Cost Virtual Reality System for Home Based Rehabilitation of the Upper Limb Following Stroke
Acronym: WiiSTAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham Trent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10057
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Virtual Reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The virtual glove in their homes for a period of 8 weeks and advised to try to build up to using the system for a maximum of 20 minutes 3 times a day for 8 weeks.
  Interventions: Device: Virtual glove
- Control (No Intervention): Usual care

INTERVENTIONS:
Device: Virtual glove — The intervention (the virtual glove) consists of a hand-mounted power unit, with four infra- red light emitting diodes (LEDs) mounted on the user's finger tips. The LEDs are tracked using one or two Nintendo Wii motes mounted by the computer screen on which the games are displayed to translate the location of the user's hand, fingers and thumb in 3D space. Three games have been produced especially for the project with the help of therapists and stroke patients. In order to play them, users have to perform the movements of reach to grasp, grasp and release, pronation and supination that are necessary to effect many activities of daily living.
  Arms: Intervention

SUMMARY:
Stroke is the third most common cause of mortality and the leading cause of long term disability worldwide with over 900,000 people living in England who have had a stroke. 75% of survivors regain their ability to walk again, however it is estimated that between 55 and 75% fail to regain satisfactory use of their impaired arm. This limits the person's independence, ability to care for themselves and reduces their quality of life. Research indicates that for optimal recovery, high levels of rehabilitation are required yet current provision often fails to meet the required levels of intensity and duration of therapy.

In conjunction with stroke patients, their families and therapists, the team developed a low cost system (the virtual glove) to encourage stroke survivors to practice arm exercises at home. The system tracks infrared light emitting diodes (LEDs) positioned on the fingers turning the hand into a game controller to play games that encourage the movements of reach, grasp and release that underlie activities of daily living.

Before examining its effectiveness, the purpose of the registered study is to determine how feasible a large trial would be in terms of whether sufficient participants could be recruited, whether they would use the glove and whether outcome measures could be collected.

Patients will be recruited if they are aged 18 years or over, are recovering from a stroke, no longer receive any other intensive rehabilitation but still experiencing difficulty using their arm. After baseline measures are collected they will be randomly allocated to either the intervention group or a control group. The intervention group will have the virtual glove and games at home for a period of eight weeks and be advised to use the equipment for 20 minutes, three times a day. The control group will continue to have whatever care they are already receiving but no new interventions.

Outcome measures will be collected at baseline, four weeks and after the equipment has been removed from their home. Outcome measures will include tests of arm function as well participant reports of how often they are using their affected arm and how easy they find activities of daily living. The therapists collecting the outcome measures will not know to which group the participants have been allocated.

Once all outcome measures are collected the two groups will be compared on how much their final outcome measures differ from those collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of stroke, no longer receiving any other intensive rehabilitation (intermediate care, early supported discharge) still experiencing residual upper limb dysfunction.

Exclusion Criteria:

* no detectable movement in the upper limb; premorbid disability in upper limb function; severe symptomatic arm or shoulder pain; severe visual impairments; other neurological illnesses such as head injury or multiple sclerosis; unstable medical condition; psychiatric illness; epilepsy triggered by screen images; cardiac pacemaker; unable to tolerate sitting in a chair for 30 minutes or follow a two stage command or living in a care home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test change from baseline at 4 weeks and 8 weeks | Baseline, 4 weeks and 8 weeks
  Change from baseline to 4 weeks and from baseline to 8 weeks in the Wolf Motor Function Test

SECONDARY OUTCOMES:
Nine-Hole Peg Test | Baseline, 4 weeks and 8 weeks

OTHER OUTCOMES:
Motor Activity Log | Baseline, 4 weeks and 8 weeks
Nottingham Extended Activities of Daily Living Scale | Baseline, 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marion Walker, PhD, Study Director — University of Nottingham